CLINICAL TRIAL: NCT02523053
Title: A Randomized Controlled Study on the Effect of Intraoperative Controlled Release 5-Fluorouracil Therapy on Anti-tumor Recurrence in Hepatocellular Carcinoma Patients With High Risk of Microvascular Invasion Presence
Brief Title: Effect of Intraoperative Controlled Release 5-Fluorouracil Therapy on Recurrence in Hepatocellular Carcinoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, Vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EHBHKY2015-01-011
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma; Recurrence
Keywords: Hepatocellular Carcinoma; Recurrence; Microvascular Invasion; 5-Fluorouracil
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Hepatectomy; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hepatectomy (Active Comparator): Surgical removal of all lesions
  Interventions: Procedure: Hepatectomy
- Hepatectomy plus 5-Fluorouracil (Experimental): Surgical removal of all lesions and intraoperative controlled release 5-Fluorouracil therapy
  Interventions: Procedure: Hepatectomy; Drug: 5-Fluorouracil

INTERVENTIONS:
Procedure: Hepatectomy — Surgical removal of all lesions
Drug: 5-Fluorouracil — Surgical removal of all lesions and intraoperative controlled release 5-Fluorouracil therapy
  Arms: Hepatectomy plus 5-Fluorouracil

SUMMARY:
The aim of this study is to confirmed the role of intraoperative controlled release 5-Fluorouracil therapy in the prevention of recurrence after surgery for HCC patients with high risk of preoperative prediction of microvascular invasion.

DETAILED DESCRIPTION:
Surgical resection is the major curative treatment for patients with hepatocellular carcinoma (HCC). However, the postoperative 5-year recurrence rate after surgical resection was significantly high, which has been reported to 40%-70%.

Recurrence after surgery is the main factor affecting the efficacy of management of hepatocellular carcinoma, however, there are few methods for the prevention of recurrence and no standard treatment for recurrent HCC following curative-intent initial surgery has been established so far. The effective prevention of recurrence is the key to improve the management of HCC.

Previous studies showed the prevalence of microvascular invasion (MVI) in one of the critical and negative prognostic factors for HCC patients after partial hepatectomy or liver transplantation. For the early stage HCC patients, preoperative prediction of MVI is helpful to identify the appropriate object of anti-recurrence treatment before or after operation.

Our another previous study established a nomogram for MVI prediction of early HCC patients, which can preoperative efficiently predict the occurrence of MVI within Milan criteria, has been published online in JAMA surgery. On the other hand, there are only few studies reported the use of controlled release 5-Fluorouracil in the treatment of digestive tract tumors.

The action time of the controlled release 5-Fluorouracil particles is more than 15 days, the diffusion radius is 4-6cm. In theory, during the operation, the drug can be given to any location that may have tumor residues, timely and conveniently, and has a long time to maintain a high drug concentration, which is conducive to kill small metastatic foci caused by MVI. However, to our best knowledge, there is no evidence of high levels of evidence-based medical evidence to confirm the value of controlled release 5-Fluorouracil in the prevention of HCC recurrence.

In view of this, we aim to implement a randomized controlled study to confirmed the role of intraoperative controlled release 5-Fluorouracil therapy in the prevention of recurrence after surgery for HCC patients with high risk of preoperative prediction of microvascular invasion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years and <=70 years of age
2. Patients preoperatively diagnosed of hepatocellular carcinoma according to the criteria of American Association for the Study of Liver Diseases(AASLD)
3. Within Milan criteria
4. Nomogram score for MVI prediction >200
5. Preoperative ECOG criteria score of 0-1
6. Child-Pugh class A liver function
7. No Anticancer treatment before surgery

Exclusion Criteria:

1. Major portal/hepatic vein invasion
2. Extrahepatic metastasis
3. Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction,which may affect the treatment of liver cancer
4. Lost to follow-up
5. Patients participating in other clinical trials
6. Patients refused to join our trial
7. Pregnant and breast-feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Time to tumor recurrence | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, MD, Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China